CLINICAL TRIAL: NCT06626516
Title: A Phase I/II Study of Tebentafusp-tebn in Combination With Liver-Directed Therapies for the Treatment of Metastatic Uveal Melanoma
Brief Title: Tebentafusp-tebn With LDT in Metastatic UM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-3117; JT 31444 (Other: JeffTrial Number)
Record Dates: First submitted 2024-09-19; First posted 2024-10-04 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Uveal Melanoma
Keywords: Uveal; uveal melanoma; metastatic uveal melanoma; melanoma; Liver-directed therapy; Liver-directed; Liver; liver-directed therapies; MUM; LDT
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Carmustine

STUDY DESIGN:
Intervention Model Description: Part 1A: Single-arm combination therapy (tebentafusp-tebn with hepatic IE with GM-CSF), with the first cohort of six patients being enrolled in a safety lead in.
  Part 1B: If the safety and preliminary efficacy in Part 1A are met, we will then proceed with a randomized phase II trial. 52 patients will be randomized in a 2:1 ratio to receive tebentafusp-tebn in combination with hepatic IE or tebentafusp-tebn alone Part 2: Single-arm, two-stage phase II trial of sequential TACE with BCNU followed by tebentafusp-tebn in 39 patients with higher liver tumor burden
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1A: Safety Lead-in (Experimental): Phase I safety lead-in followed by a phase II trial with 6-month PFS rate as the preliminary efficacy endpoint.
  All patients will receive a 4-week induction course of tebentafusp-tebn alone (Cycle 1) using the approved step-up dosing regimen. Should the 4th dose be tolerated well as an outpatient, patients will receive their first IE treatment on Cycle 2 week 1 followed by continued weekly tebentafusp-tebn on weeks 2, 3, and 4 of Cycle 2 (See Figure 1). Patients will not receive tebentafusp-tebn concurrently with their first IE treatment during Week 1 of Cycle 2. Should Cycle 2 be well tolerated, patients may receive both tebentafusp-tebn and IE on Week 1 of subsequent
  Interventions: Drug: Tebentafusp-Tebn; Drug: GM-CSF (Sargramostim)
- Part 1B: Combination (Active Comparator): If the safety and preliminary efficacy in Part 1A are met, we will then proceed with a randomized phase II trial.
  52 patients will be randomized in a 2:1 ratio to receive tebentafusp-tebn in combination with hepatic IE or tebentafusp-tebn alone, with PFS as the primary endpoint. Patients randomized to tebentafusp-tebn + IE arm will be treated as Part 1A.
  Interventions: Drug: Tebentafusp-Tebn; Drug: GM-CSF (Sargramostim)
- Part 1B: Tebentafusp-tebn alone (Active Comparator): If the safety and preliminary efficacy in Part 1A are met, we will then proceed with a randomized phase II trial.
  52 patients will be randomized in a 2:1 ratio to receive tebentafusp-tebn in combination with hepatic IE or tebentafusp-tebn alone, with PFS as the primary endpoint. Patients randomized to tebentafusp-tebn alone will receive weekly treatment using the approved step-up dosing regimen.
  Interventions: Drug: Tebentafusp-Tebn
- Part 2: Efficacy of Combo (Active Comparator): To assess the efficacy of tebentafusp-tebn in sequence with TACE in HLA-A*0201-positive patients with metastatic uveal melanoma to the liver
  Interventions: Drug: Tebentafusp-Tebn; Drug: BCNU

INTERVENTIONS:
Drug: Tebentafusp-Tebn — Dosing: All patients enrolled in this study will receive treatment with tebentafusp-tebn based on the approved step-up dosing regimen of 20 mcg on C1D1, 30 mcg on C1D8, then 68 mcg weekly beginning on C1D15 and thereafter. This escalated dose administered at C1D15 will be the dose used for the remainder of the treatment period unless dose reduction is implemented for toxicity. Beginning with C1D8, tebentafusp-tebn will be administered on the scheduled day (± 2 days), and consecutive infusions of tebentafusp-tebn must be administered at least 5 days apart.
  Other Names: kimmtrak; IMCgp100
Drug: GM-CSF (Sargramostim) — Recombinant human GM-CSF (Sargramostim, Leukine®, Sanofi US) 1,500mg will be mixed with ethiodized oil (Ethiodol®). The GM-CSF/ethiodized oil mixture will be injected selectively into one of the hepatic lobes, followed by infusion of gelatin sponge particles to achieve the stasis of blood flow. This will repeat every 4 weeks.
  Other Names: yeast-derived recombinant human GM-CSF; Leukine; Hepatic Immunoembolization; GM-CSF; Sargramostim
  Arms: Part 1A: Safety Lead-in; Part 1B: Combination
Drug: BCNU — Patients will be treated with hepatic artery infusion of 300mg BCNU (1,3-bis [2-chloroethyl]-1-nitrosourea, Carmustine) dissolved in ethiodized oil followed by embolization with gelatin sponge particles [TACE with BCNU 300mg]; every 4 weeks +/- 7 days in the case of either bilobar or unilobar metastasis
  Other Names: Carmustine; BiCNU; bis-chloroethylnitrosourea; Hepatic Chemoembolization; 1,3-bis [2-chloroethyl]-1-nitrosourea
  Arms: Part 2: Efficacy of Combo

SUMMARY:
This study is a multicenter, open label phase I/ II trial to assess the safety and clinical efficacy of tebentafusp-tebn in combination with liver-directed therapies in HLA-A*0201 positive patients with metastatic uveal melanoma. In Part 1 of the study, the Prinicipal Investigator will investigate the safety and efficacy of tebentafusp-tebn in combination with hepatic IE in patients with a low to moderate hepatic disease burden. In Part 2, the study will investigate the efficacy of tebentafusp-tebn in combination with TACE in patients with bulky hepatic disease.

DETAILED DESCRIPTION:
PART 1: TEBENTAFUSP AND IE Part 1A, Phase I/II: This is a single-arm study of 18 patients treated with combination therapy (tebentafusp-tebn with hepatic IE with GM-CSF), with the first cohort of six patients being enrolled in a safety lead in. The SKCC DSMC will monitor and approve the cohort expansion, please refer to section 3.2 for further details. The preliminary clinical efficacy endpoint is defined as a target 6-month liver-specific PFS rate of 60%. All patients will receive a 4-week induction course of tebentafusp-tebn alone (Cycle 1) using the approved step-up dosing regimen. Should the 4th dose be tolerated well as an outpatient, patients will receive their first IE treatment on Cycle 2 week 1 followed by continued weekly tebentafusp-tebn on weeks 2, 3, and 4 of Cycle 2 (See Figure 1). Patients will not receive tebentafusp-tebn concurrently with their first IE treatment during Week 1 of Cycle 2. Should Cycle 2 be well tolerated, patients may receive both tebentafusp-tebn and IE on Week 1 of subsequent cycles, with tebentafusp administered alone on weeks 2-4 of subsequent cycles.

Part 1B, Phase II: If the safety and preliminary efficacy in Part 1A are met, the study will then proceed with a randomized phase II trial. 52 patients will be randomized in a 2:1 ratio to receive tebentafusp-tebn in combination with hepatic IE or tebentafusp-tebn alone, with PFS as the primary endpoint. Secondary endpoints will include ORR, duration of response, systemic PFS, and OS. Patients randomized to tebentafusp-tebn + IE arm will be treated as above (See Figure 1). Patients randomized to tebentafusp-tebn alone will receive weekly treatment using the approved step-up dosing regimen. Tumor biopsies will be optional for all patients on this portion of the study; however, peripheral blood and ctDNA will be collected as above.

PART 2: TEBENTAFUSP AND TACE The trial will conduct a single-arm, two-stage phase II trial of sequential TACE with BCNU followed by tebentafusp-tebn in 39 patients with higher liver tumor burden (greatest tumor size >5 cm and/or ≥50% liver involvement on imaging). Patients with unilobar disease will first receive at least two treatments of TACE with 300mg BCNU (Cycles 1-2, See Figure 2A); patients with bilobar disease will receive at least 4 treatments (Cycles 1-4, See Figure 2B). Following completion of the TACE course, patients will receive tebentafusp-tebn on a weekly basis at the approved step-up dosing regimen.

Patients will undergo imaging studies at baseline, after completion of every two TACE treatments, and every 8 weeks thereafter while on tebentafusp-tebn alone. Tumor biopsies will be performed at baseline, following TACE, and after 4 weeks of treatment with tebentafusp-tebn. Peripheral blood will be collected for serum cytokine and PBMC analysis after completion of each TACE treatment and every 4 weeks thereafter. ctDNA will be collected at the time of each interval scan. Correlative studies will be performed as above in Part 1. Following the initial TACE treatments and subsequent tebentafusp induction, patients may receive additional TACE treatments at the discretion of the investigator. These will only be offered once a patient is through tebentafusp induction and has transitioned outpatient. Patients who proceed with additional TACE will hold tebentafusp the week of treatment and be followed with weekly labs to ensure return to baseline before proceeding with next scheduled tebentafusp at the discretion of the investigator.

Participants will continue treatment until confirmed disease progression, or for as long as the patient is deriving clinical benefit in the opinion of the treating investigator with approval of the study PI. The treating investigator may provide rationale and request approval for treatment beyond progression via email to the Study PI.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years of age 2. Histologically or cytologically confirmed metastatic uveal melanoma in the liver. Patients must have at least one measurable liver metastasis that is ≥ 10 mm in longest diameter by CT scan or MRI. Extra-hepatic disease is allowed. 3. Tumor Size Criteria: i. Part 1: Total volume of tumor must be < 50% of the liver involvement by CT or MRI; M1a or M1b disease with largest tumor ≤ 5 cm ii. Part 2: M1b disease with largest tumor > 5 cm, M1c disease, or ≥ 50% liver involvement by CT or MRI 4. No prior systemic treatment with tebentafusp-tebn 5. Prior therapy: i. Part 1: Patients must be treatment naïve in the metastatic setting.

1. Prior surgery or ablation for oligometastatic disease is allowable.
2. Palliative radiation of non-target lesions also allowable. ii. Part 2: Patients may have had prior systemic therapy with chemotherapy, immunotherapy, or targeted therapy. They can also have had prior liver directed therapy including surgery, ablation, immunoembolization, or radioembolization. However cannot have had more than two prior lines of treatment total.

6. HLA-A*0201 positive 7. ECOG performance status or 0 or 1 at the time of screening 8. Life expectancy of greater than 3 months as assessed by the investigator 9. Patients must have normal organ and bone marrow function as defined below:

1. Platelet count ≥ 100,000/mm³
2. Hemoglobin > 8.0g/dL
3. ANC ≥ 1500
4. AST and/or ALT < 3x upper limited of normal (ULN)
5. Total bilirubin ≤ 2.0 mg/ml
6. Note: Patients with hyperbilirubinemia clinically consistent with an inherited disorder of bilirubin metabolism (e.g., Gilbert syndrome) will be eligible at the discretion of the treating physician and/or the principal investigator.
7. PT/PTT < 1.5x ULN
8. Creatinine clearance > 60mL/min
9. Potassium, magnesium, corrected calcium, and phosphate within normal laboratory parameters 10. Women must not be pregnant or breast-feeding. 11. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for the 6 months after the final dose of the study drug. Women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

   12. Male patients treated or enrolled on this protocol must be surgically sterile or use double barrier contraception methods from enrollment through treatment, and for 6 months after completion of study therapy.

   13. Ability to understand and the willingness to sign a written informed consent document.

4.1.2 Exclusion Criteria

1. Parts 1 and 2:

   1. Failure to meet any of the criteria set forth in the Inclusion criteria section
   2. History of prior tebentafusp-tebn use
   3. Prior chemoembolization in Part 2 is not permitted
   4. History of severe immediate or delayed hypersensitivity reaction to biologic drugs, monoclonal antibodies, iodinated contrast agent
   5. Presence of symptomatic liver failure including ascites and hepatic encephalopathy
   6. Presence of symptomatic or untreated central nervous system (CNS) metastases, or CNS metastases that require corticosteroids within 21 days prior to initiation of study therapy. Patients with brain metastases may be eligible if lesions have been treated with local therapy and there is no evidence of CNS disease progression for at least 4 weeks as measured by MRI prior to first dose of study drug
   7. History of another malignancy except for: 1) those who have been disease-free for 3 years prior to study treatment; 2) patients with a history of completely resected non-melanoma skin cancer; 3) patients with indolent secondary malignancies not requiring active therapy; 4) patients with completely resected carcinoma in situ. Consult the study Principal Investigator if unsure whether second malignancies meet the requirements specified above.
   8. Major surgery within 2 weeks of the first dose of study drug (minimally invasive procedures such as bronchoscopy, tumor biopsy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery and are not exclusionary)
   9. Radiotherapy within 2 weeks of the first dose of study drug, with the exception of palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass
   10. No outstanding toxicities from prior therapies greater than Grade 1. Except for prior immune related side effects such as endocrinopathy that are managed with a stable dose of thyroid or steroid supplement.
   11. Use of any investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of study therapy and during the study.
   12. Use of hematopoietic colony-stimulating growth factors (eg. G-CSF, GMCSF, M-CSF) within 14 days prior to study treatment initiation. An erythroid-stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment and the patient is not red blood cell transfusion dependent.
   13. Known history of human immunodeficiency virus infection (HIV). Testing for HIV is not necessary unless clinically indicated
   14. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Testing for HBV or HCV status is not necessary unless clinically indicated or if the patient has a history of HBV or HCV infection.
   15. Patients receiving systemic steroid therapy or any immunosuppressive medication. Local steroid therapies (eg, otic, ophthalmic, intra-articular or inhaled medications) are acceptable.
   16. History of bleeding diathesis
   17. Pregnant, likely to become pregnant, or breastfeeding women
   18. Uncontrolled concurrent illness, evaluated at investigator discretion
   19. Biliary obstruction, biliary stent or prior biliary surgery except cholecystectomy, or any anatomic abnormalities that would interfere with immunoembolization or chemoembolization:
   20. Patients with occlusion of the main portal vein
   21. Inadequate collateral flow around an occluded portal vein as determined by angiography
   22. Arteriovenous shunt identified on arteriography of the hepatic artery
   23. Any medical condition that, in the Investigator's judgement, would prevent patient participation in the clinical study due to safety concerns, compliance with study procedures or interpretation of study results
2. Part 1 Only:

   1. History of severe immediate or delayed hypersensitivity reaction to GM-CSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Part 1A: Safety lead-in | From when the patient receives the first study treatment to 7 days (for non-serious AEs) or 30 days (for SAEs) after completion of study treatment or withdrawal from the study.
  Adverse events (AEs) according to NCI CTCAE Version 5.0. Safety and tolerability data will be presented by treatment arm using the safety population. Safety data will be summarized descriptively and will not be formally analyzed. AE presentation will include incidence, severity, and relationship to study drug.
Part 1A: Efficacy | From when the patient receives the first study treatment to 6 months after first treatment
  6-month progression-free survival rate as determined by response criteria (RECIST 1.1). Will be summarized by count and percentage along with the two-sided 90% exact confidence interval (CI).
Part 1B: Progression-free Survival | From when patient joins study until disease progression or death, up to 2.5 years after last patient's last treatment.
  Defined as the time from the date of randomization until the date of objective disease progression or death by any cause. The primary Progression-free Survival (PSF) analysis will use a one-sided log-rank test, with a type I error of 0.05. In addition, PFS will be analyzed using Cox proportional hazards model and the estimated HR with 90% Confidence Interval (CI) will be reported. Kaplan-Meier curves of PFS will be presented by treatment arm along with estimated medians PFS (CIs).
Part 2: 6-month progression-free survival rate | From when the patient receives the first study treatment to 6 months after first treatment.
  As determined by response criteria (RECIST 1.1). Defined as the proportion of patients alive and progression-free at 6 months after treatment initiation. Will be summarized by count and percentage. In addition, a two-sided 90% Confidence Interval (CI) based on the method of Koyama and Chen will be provided. This method is appropriate because it is proposed for Simon's 2-stage design, accounting for the inherent futility analysis.

SECONDARY OUTCOMES:
All toxicities using the NCI CTCAE Version 5.0 | From when the patient receives the first study treatment to 7 days (for non-serious AEs) or 30 days (for SAEs) after completion of study treatment or withdrawal from the study.
  Safety and tolerability data will be presented by treatment arm using the safety population. Safety data will be summarized descriptively and will not be formally analyzed. AE presentation will include incidence, severity, and relationship to study drug.
Overall response rate (ORR) | From when the patient receives the first study treatment to at least one year (and up to 2.5 years) after discontinuing treatment
  Count and percentage of patients with a tumor response (Complete Response/Partial Response)
Liver-specific progression-free survival | From when patient joins study until disease progression or death, up to 2.5 years after last patient's last treatment.
  As determined by response criteria (RECIST 1.1). Defined as the proportion of patients alive and progression-free at 6 months after treatment initiation. Will be summarized by count and percentage.
Overall survival | From the start of the treatment to death due to any cause (assessed up to 2.5 years after last patient's last treatment)
  Measured from the start of the treatment to death due to any cause. Date and cause of death will be recorded. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive. The cause of death will be categorized as either cancer-related or cancer-unrelated.

CONTACTS AND LOCATIONS:
Overall Officials: Rino Seedor, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No